CLINICAL TRIAL: NCT05698667
Title: Surgeon-performed Outpatient Transoral and Transcervical Ultrasound for the Diagnostic Work-up of Oropharynx Cancer: a Feasibility Study
Brief Title: Outpatient Ultrasound for the Diagnostic Work-up of Oropharynx Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Novo Nordic Foundation (Other)
Responsible Party: Principal Investigator, Martin Garset-Zamani, MD, Principal Investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Transoral US Feasibility
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Oropharynx Cancer; Oropharynx Neoplasm; Tonsil Cancer; Tonsil Neoplasm; Tonsil Hypertrophy; Tonsil Lymphoma; Base of Tongue Tumor; Base of Tongue Carcinoma
MeSH Terms: conditions — Oropharyngeal Neoplasms; Tonsillar Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oropharynx Ultrasound (Experimental): Transoral and transcervical ultrasound of the oropharynx, including the tonsils and tongue base.
  Interventions: Diagnostic Test: Transoral ultrasound; Diagnostic Test: Transcervical ultrasound

INTERVENTIONS:
Diagnostic Test: Transoral ultrasound — Under local anesthetic with xylocaine spray in the oropharynx, the tonsils and tongue base are scanned with small-footprint, high-frequency ultrasound transducers (such as the 18XL5s hockey-stick from BK Medical)
Diagnostic Test: Transcervical ultrasound — The tongue base and tonsils are scanned externally via the neck, where a (preferably low-frequency) transducer is placed onto the skin above the hyoid bone to visualize the tongue base. The tonsils are visualized adjacent to the tongue base on either side and are located deep to the submandibular glands in a oblique coronal plane.

SUMMARY:
The aim of the study was to examine the detection rate and tumor size evaluation in patients with suspected oropharynx cancer using a new technique with transoral ultrasound of the oropharynx. The new technique was compared to Magnetic Resonance Imaging (MRI). The study investigators included patients referred to a tertiary head & neck cancer center in Copenhagen, Denmark, with suspicion of oropharynx cancer. Patients supplied written informed consent and were included and ultrasound scanned with local anesthesia in the outpatient clinic. Blinded assessment of MRI's was performed for tumor detection and compared to ultrasound with the reference standard being histopathology biopsy results.

DETAILED DESCRIPTION:
An explorative diagnostic study was performed at the Department of Otorhinolaryngology, Head & Neck Surgery, Copenhagen University Hospital - Rigshospitalet, Denmark from October 1st, 2021, to April 30th, 2022. The study investigators invited adult patients from the outpatient cancer clinic referred with a suspicion of oropharynx cancer to participate in the study. At the study investigators' center, all head & neck cancer patients receive diagnostic work-up which includes clinical exam, flexible laryngoscopy with narrow-band imaging, surgeon-performed neck ultrasound and biopsy and/or cytology with same-day results. Patients were enrolled after verbal and written consent and were offered an ultrasound examination of the oropharynx as an addition to the standard diagnostic workup in the outpatient clinic. All included patients also received an MRI of the head and neck. Clinical data including age, sex, smoking habits, alcohol consumption, date of MRI scan, and histopathology results were obtained from medical charts after inclusion.

Interventions included transoral ultrasound of the tonsils and base of tongue, conducted with BK5000 ultrasound machines using the X18L5s "hockey stick" transducer. Transcervical ultrasound was also performed in patients where a tongue base cancer was most likely. Standard linear neck transducers (X18L5) or a curved 9C2 transducer was used. The tonsils and tongue base were scanned in two planes if possible, and doppler flow was recorded as well. Ultrasound images were stored as video clips.

The detection of tumors with ultrasound was recorded as "positive" if a well-defined tumor was seen that was clearly visualized compared to the contralateral side. A "negative" result was given if no tumors were suspected on either side. An "inconclusive" result was given if a tumor was not clear, but there was suspicious asymmetry visualized. The anatomical sub-location of tumors were stratified into right and left tonsil, tongue base, overlapping tonsil and tongue base, and "other" sub-locations. "Other" sub-locations included the soft palate, uvula, oropharynx posterior wall, vallecula, anterior pharyngeal arch and posterior pharyngeal arch.

MRI was used as the reference test. An expert neuroradiologist blinded to ultrasound results and histopathology rated all tests for tumor detection in the oropharynx and tumor size in detected tumors.

Statistical analysis:

Tumor detection of oropharynx ultrasound and MRI will be compared using the histopathologic diagnosis (cancer or benign) as reference standard to calculate sensitivity, specificity, positive- and negative predictive values (PPV, NPV).

Inconclusive tests will be analyzed as a positive result due to the clinical consequences often leading to diagnostic tonsillectomy.

McNemar's test for differences between sensitivity, specificity, PPV and NPV between ultrasound and MRI will be calculated.

The greatest tumor diameter will be compared between ultrasound and MRI using scatter plots and the Pearson's R correlation coefficient. Tumor volumes calculated using the formula for an ellipse: π/6 * craniocaudal * anteroposterior * mediolateral will be compared. Statistical analysis will be performed using R software version 4.2.2.

ELIGIBILITY:
Inclusion Criteria (any of the following):

* Visible and/or palpable tumor or asymmetry of the tonsils, tongue base or oropharynx.
* Subjective symptoms of oropharynx cancer including dysphagia, odynophagia and/or referred otalgia.

Exclusion Criteria:

* Unable to understand Danish or English.
* Unable to provide written informed consent.
* Age younger than 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with oropharynx cancer detected by ultrasound compared to MRI | Within two weeks.
  Patients with cancer (histopathology verified) correctly detected by a positive ultrasound or MRI test result.

SECONDARY OUTCOMES:
Greatest tumor diameter compared between ultrasound and MRI. | 1 day
  Greatest tumor diameter measured in millimeters.
Proportion of patients without oropharynx cancer detected by ultrasound compared to MRI | Within three months.
  Patients with benign tonsillar asymmetry (histopathology verified) correctly detected by a negative ultrasound or MRI test result.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Todsen, MD, PhD, Study Director — Rigshospitalet, Denmark
Locations (1):
- Department of Otorhinolaryngology, Head & Neck Surgery & Audiology, Copenhagen, Denmark